CLINICAL TRIAL: NCT04242277
Title: A Prospective, Multi-center, Randomized, Double-arm Trial to Determine the Impact of the SELENE System on Positive Margin Rates in Breast Conservation Surgery.
Brief Title: Wide-field Optical Coherence Tomography Imaging of Excised Breast Tissue.
Status: Completed | Type: Observational
Sponsor: Perimeter Medical Imaging (Industry)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: PER-19-03
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- WF-OCT imaging of excised breast lumpectomy tissue: Excised lumpectomy tissue from all consented patients will be imaged on an investigational OCT-based device. No clinical decisions will be made based on the images acquired.
  Interventions: Device: Investigational WF-OCT device

INTERVENTIONS:
Device: Investigational WF-OCT device — Excised lumpectomy tissue will be imaged on an investigational WF-OCT device

SUMMARY:
This is a single-arm, multi-center data collection study designed to collect WF-OCT imaging data of excised breast tissue margins with corresponding margin status from histopathology.

DETAILED DESCRIPTION:
Data collected during this study will be used for product development by the study sponsor, Perimeter Medical Imaging.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* Invasive ductal breast carcinoma and ductal carcinoma in situ having undergone breast conservation surgery
* May include neo-adjuvant treated subjects (chemotherapeutic, endocrine therapy, or radiation)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Metastatic cancer (Stage IV)
* Lobular carcinoma as primary diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Consented patients meeting eligibility criteria, undergoing breast conservation surgery.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
WF-OCT image acquisition of excised lumpectomy tissue margins | 1 year
  This is a data collection study. The primary outcome is the collection of WF-OCT images of excised lumpectomy tissue margins.

CONTACTS AND LOCATIONS:
Overall Officials: Savitri Krishnamurthy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided